CLINICAL TRIAL: NCT01540253
Title: A Phase I Study of the PI3-Kinase Inhibitor BKM120 in Combination With Docetaxel in Patients With Advanced Solid Tumors.
Brief Title: PI3K Inhibitor BKM120 and Docetaxel in Treating Patients With Advanced Solid Tumor That is Locally Advanced, Cannot Be Removed By Surgery, or Metastatic
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 186510; NCI-2011-00521 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 186510 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2011-11-29; First posted 2012-02-28 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — NVP-BKM120; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (enzyme inhibitor and chemotherapy) (Experimental): Patients receive PI3K inhibitor BKM120 PO QD and docetaxel IV over 1 hour on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: PI3K inhibitor BKM120; Drug: docetaxel; Other: pharmacological study; Other: questionnaire administration; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: PI3K inhibitor BKM120 — Given PO
  Other Names: BKM120; PI3K_Inhibitor_BKM120
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: questionnaire administration — Ancillary studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of PI3K inhibitor BKM120 when given together with docetaxel in treating patients with advanced solid tumor that is locally advanced, cannot be removed by surgery, or metastatic. PI3K inhibitor BKM120 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving PI3K inhibitor BKM120 together with docetaxel may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the dose-limiting toxicities and identify the recommended phase II dose of the combination of docetaxel and BKM 120 (P13K inhibitor BKM120) in patients with advanced solid tumors.

II. To determine the safety and tolerability of this combination. III. To determine any pharmacokinetic (PK) interaction between BKM12O and docetaxel.

SECONDARY OBJECTIVES:

I. To assess any preliminary evidence of efficacy with this combination in patients with advanced cancers.

II. To evaluate phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha (PIK3CA) mutations as predictive biomarkers of efficacy for the combination.

III. To evaluate PIK3CA polymorphisms and polymorphisms in BKM120 transport and metabolism as predictors of toxicity and/or efficacy.

OUTLINE: This is a dose-escalation study of PI3K inhibitor BKM120.

Patients receive PI3K inhibitor BKM120 orally (PO) once daily (QD) and docetaxel intravenously (IV) over 1 hour on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent granted prior to initiation of any study-specific screening procedures, given with the understanding that the patient has the right to withdraw from the study at any time, without prejudice
* Histologically or cytologically confirmed diagnosis of solid malignancy; patient should have locally advanced, inoperable or metastatic solid tumor with at least one site of measurable disease [if applicable] (per Response Evaluation Criteria in Solid Tumors [RECIST] for solid tumors or the appropriate disease classification/criteria for the target population)
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Life expectancy of >= 12 weeks
* Platelet count >= 100 x 10^9/L
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Hemoglobin (Hgb) >= 9 gm/dl
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) within upper limits of normal (ULN) range (or =< 3.0 x ULN if liver metastases are present)
* Serum bilirubin within ULN range (or =< 1.5 x ULN if liver metastases are present; or total =< 3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert syndrome)
* Serum creatinine =< 1.5 x ULN or 24-hour clearance >= 50 mL/min
* Serum amylase =< ULN
* Serum lipase =< ULN
* Fasting plasma glucose =< 120 mg/dl
* International normalized ratio (INR) =< 2
* Magnesium >= the lower limit of normal
* Potassium within normal limits
* Total calcium (corrected for serum albumin) within normal limits (bisphosphonate use for malignant hypercalcemia control is not allowed)
* Women of childbearing potential must have a negative pregnancy test performed within 48 hours prior to the start of study drug
* Male and female subjects of child-bearing potential must agree to use double-barrier contraceptive measures, oral contraception, or avoidance of intercourse during the study and for 90 days after last investigational drug dose received

Exclusion Criteria:

* Previous anti-cancer chemotherapy, immunotherapy or investigational agents < 4 weeks prior to the first day of study defined treatment; palliative radiation < 2 weeks; patients who receive gamma knife radiosurgery for brain metastases are eligible if procedure was performed > 4 weeks before treatment is started, is clinically stable and has been on stable low dose corticosteroid treatment (e.g. dexamethasone 2 mg/day, prednisolone 10 mg/day for at least 14 days before start of study treatment are eligible); ongoing hormonal therapies (luteinizing hormone-releasing hormone [LHRH] antagonists, megestrol) are allowed
* Previous treatment with a phosphatidylinositol 3-kinase (P1-3K) inhibitor
* Patients with a known hypersensitivity to BKM120 or to its excipients
* Patients with acute or chronic liver, renal disease or pancreatitis
* Patients have any of the following mood disorders as judged by the investigator or a psychiatrist, or who meets the cut-off score of >= 12 in the Patient Health Questionnaire (PHQ-9) or a cut-off of >= 15 in the Generalized Anxiety Disorder (GAD-7) mood scale, respectively, or selects a positive response of '1, 2, or 3' to questions number 9 regarding potential for suicidal thoughts in the PHQ-9 (independent of the total score of the PHQ-9)

  * Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others)
  * >= Common Terminology Criteria for Adverse Events (CTCAE) grade 3 anxiety
* Patients with diarrhea >= CTCAE grade 2
* Patient has active cardiac disease including any of the following:

  * Left ventricular ejection fraction (LVEF) < 50% as determined by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO)
  * Corrected QT interval (QTc) > 480 msec on screening electrocardiogram (ECG) (using the QT interval corrected for Fridericia [QTcF] formula)
  * Angina pectoris that requires the use of anti-anginal medication
  * Ventricular arrhythmias except for benign premature ventricular contractions
  * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication
  * Conduction abnormality requiring a pacemaker
  * Valvular disease with document compromise in cardiac function
  * Symptomatic pericarditis
  * Previous history of QTc prolongation as a result of other medication that required discontinuation of that medication
  * Congenital long QT syndrome or 1st degree relative with unexplained sudden death under 40 years of age
* Patient has a history of cardiac dysfunction including any of the following:

  * Myocardial infarction within the last 6 months, documents by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function
  * History of documents congestive heart failure (New York Heart Association functional classification III-IV)
  * Documented cardiomyopathy
* Active clinically serious infections defined as >= grade 2 according to National Cancer Institute (NCI) CTCAE, version 4.0
* Substance abuse, medical, psychological or social conditions that may, in the opinion of the Investigator, interfere with the patient's participation in the study or evaluation of the study results
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her protocol compliance
* Patient has poorly controlled diabetes mellitus, steroid-induced diabetes mellitus, or glycosylated hemoglobin (HbA1c) > 7%
* Known human immunodeficiency virus (HIV) infection
* Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol
* Significant symptomatic deterioration of lung function; if clinically indicated, pulmonary function tests including measures of predicted lung volumes, diffusion capacity of carbon monoxide (DLco), oxygen (O2) saturation at rest on room air should be considered to exclude pneumonitis or pulmonary infiltrates
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKM 120 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection); patients with unresolved diarrhea will be excluded as previously indicated
* Patients who have been treated with any hematopoietic colony-stimulating growth factors (e.g., filgrastim [G-CSF], sargramostim [GM-CSF]) =< 2 weeks prior to starting study drug; erythropoietin or darbepoetin therapy, if initiated at least 2 weeks prior to enrollment, may be continued
* Patients who have taken herbal medications and certain fruits within 7 days prior to starting study drug; herbal medications include, but are not limited to St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng; fruits include the cytochrome P450, family 3, subfamily A (CYP3A) inhibitors Seville oranges, grapefruit, pummelos, or exotic citrus fruits
* Patients who have received wide field radiotherapy =< 4 weeks or limited field radiation for palliation =< 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Women who are pregnant or breast feeding or adults of reproductive potential not employing an effective method of birth control; double barrier contraceptives must be used through the trial by both sexes; oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study; women of child-bearing potential, defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months), must have a negative serum pregnancy test =< 48 hours prior to initiating treatment
* Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum follicle-stimulating hormone (FSH) levels > 40 mlU/mL (for US only: and estradiol < 20 pg/mL) or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago; in the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during treatment for 4 weeks (5 T1/2) after stopping treatment; the highly effective contraception is defined as either:

  * True abstinence: when this is in line with the preferred and usual lifestyle of the subject; periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago; in case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate); for female subjects on the study, the vasectomized male partner should be the sole partner for that patient
  * Use of a combination of any two of the following (a+b):

    * a) Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    * b) Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
  * Oral contraception, injected or implanted hormonal methods are not allowed as BKM120 potentially decreases the effectiveness of hormonal contraceptives
  * Women of child-bearing potential must have a negative serum pregnancy test =< 48 hours prior to initiating treatment
  * Fertile males, defined as all males physiologically capable of conceiving offspring must use condom during treatment, for 4 weeks (5 T1/2) after stopping treatment and for additional 12 weeks (16 weeks in total after study drug discontinuation) and should not father a child in this period
  * Female partner of male study subject should use highly effective contraception during dosing of any study agent and for 16 weeks after final dose of study therapy
* Inability to swallow oral medications
* Significant gastrointestinal disorder, in the opinion of the investigator, could interfere with the absorption of BKMI20 (e.g. significant, uncontrolled inflammatory bowel disease, history of abdominal fistula or gastrointestinal [GI] perforation within 6 months, extensive small bowel resection and requirement for tube feeding or parenteral hydration/nutrition)
* Patients who are currently receiving treatment with medication with a known risk to prolong the QT interval or inducing Torsades de Pointes and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug
* Patients receiving chronic treatment with steroids or another immunosuppressive agent; Note: topical applications (e.g. rash), inhaled sprays (e.g. obstructive airways diseases), eye drops or local injections (e.g. intra-articular) are allowed; patients with previously treated brain metastases, who are on stable low dose corticosteroids treatment (e.g. dexamethasone 2 mg/day, prednisolone 10 mg/day) for at least 14 days before start of study treatment are eligible
* Patients who are currently treated with drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug (please note that co-treatment with weak inhibitors of CYP3A is allowed)
* Patients who have received chemotherapy or targeted anticancer therapy =< 4 weeks (6 weeks for nitrosourea, antibodies or mitomycin-C) prior to starting study drug must recover to a grade 1 before starting the trial
* Patients who have received any continuous or intermittent small molecule therapeutics (excluding monoclonal antibodies) =< 5 effective half-lives prior to starting study drug or who have not recovered from side effects of such therapy
* No concurrent intake of valproic acid, rifampin, phenobarbital, phenytoin, or carbamazepine
* Patients who are currently taking therapeutic doses of warfarin sodium or any other Coumadin derivative anticoagulant
* Patient is unable or unwilling to abide by the study protocol or cooperate fully with the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-05; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) or recommended phase 2 dose of PI3K inhibitor BKM120 | 21 days
  Adverse events (AE) will be coded and evaluated for severity using NCI CTCAE, version 4.0 and will be summarized by system organ class and preferred term.
Incidence AE and tolerability of PI3-kinase inhibitor BKM120 in combination with docetaxel | Up to 30 days after completion of treatment
  AE will be coded and evaluated for severity using NCI CTCAE, version 4.0 and will be summarized by system organ class and preferred term.

SECONDARY OUTCOMES:
Objective response rate (ORR) as assessed by the proportion of patients with a confirmed complete response (CR) or partial response (PR) | Up to 6 courses
  The ORR will be calculated as the number of patients with a confirmed complete or partial response divided by the total number of patients. Tumor response will be summarized for the evaluable patient population, and the 95% confidence interval for ORR (complete response [CR] + partial response [PR]) will be presented. Response will be evaluated by revised RECIST 1.1 criteria.
Progression-free survival (PFS) | Up to 3 years
PK parameters of PI3-kinase inhibitor BKM120 | Baseline, days 1-7 of course 1, and then day 1 of all subsequent courses

CONTACTS AND LOCATIONS:
Overall Officials: Alex Adjei, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States